CLINICAL TRIAL: NCT04772443
Title: A Randomized, Double-blind, Multi-center, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DWJ1506 and DWJ1507
Brief Title: Evaluate the Efficacy and Safety of DWJ1506 and DWJ1507
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWJ1507301
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DWJ1506 (Experimental)
  Interventions: Drug: DWJ1506
- DWJ1507 (Experimental)
  Interventions: Drug: DWJ1507
- DWC202011 (Active Comparator)
  Interventions: Drug: DWC202011
- DWJ1177 (Active Comparator)
  Interventions: Drug: DWJ1177

INTERVENTIONS:
Drug: DWJ1506 — DWJ1506
  Arms: DWJ1506
Drug: DWJ1507 — DWJ1507
  Arms: DWJ1507
Drug: DWC202011 — DWC202011
  Arms: DWC202011
Drug: DWJ1177 — DWC202011
  Arms: DWJ1177

SUMMARY:
The purpose of this study is to determine the efficacy and safety of DWJ1506 and DWJ1507 in the patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or over
2. Patients with LDL-C levels ≤ 250 mg/dL, TG < 500 mg/dL
3. Subjects who voluntarily decided to participate and provided written consent after being told of the objectives, method, and effects of this study

Exclusion Criteria:

1. Severe congestive hear failure
2. Current active liver disease
3. The use of prohibiterd concomitant therapies
4. Severe gastrointestinal diseases: active ulcer, gastrointestinal or rectal bleeding, active inflammatory bowel syndrome, biliary duct obstruction, active gastritis that is not controlled by medication, etc.

6.Women who were of childbearing potential without contraception, pregnant, or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
LDL-C levels at week 8 | Week 8
  Change from baseline in LDL-C level at week 8 after administration of the IP

IPD SHARING:
Plan to Share IPD: Yes